CLINICAL TRIAL: NCT05513716
Title: Molecular Characterisation of Colorectal Cancer Peritoneal Metastases: Genomic and Transcriptomic Analysis With Correlation of Clinical Outcomes
Brief Title: Molecular Characterisation of Colorectal Cancer Peritoneal Metastases
Acronym: COLOMET II
Status: Recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp216
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal Cancer Peritoneal Metastatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archival formalin-fixed, paraffin-embedded (FFPE) tumour tissue from colorectal cancer peritoneal metastasis and paired primary tumours, where available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Colorectal cancer patients
  Interventions: Other: Retrospective tissue sample analysis

INTERVENTIONS:
Other: Retrospective tissue sample analysis — Archival formalin-fixed, paraffin-embedded (FFPE) tumour tissue from colorectal cancer peritoneal metastasis and paired primary tumours, where available - taken as standard care

SUMMARY:
This project aims to characterise the tumour cell and tumour microenvironment of colorectal cancer peritoneal metastases, understand molecular changes leading to colorectal peritoneal metastasis, identify potential biomarkers and novel treatment strategies.

DETAILED DESCRIPTION:
The peritoneum is the second most common site for recurrence in colorectal cancer (CRC). Cancer spread to the peritoneum (colorectal cancer peritoneal metastases, CRPM) cause severe symptoms in patients and lead to shortened survival. The only definitive treatment available is a complex and aggressive surgical procedure involving radical removal of organs and the internal lining of the abdomen.

The biology of CRPM and correlations with clinical outcomes has been reported in small numbers of patients. There has been limited research on how extended cancer mutations lead to metastases and how this can affect treatment or survival. Understanding how genetic mutations evolve in CRPM and the role of the tumour microenvironment are important for optimising treatment and prevent the spread of cancer.

This study proposes completing cancer genetic profiling on archived tissue removed routinely from patients who previously have had surgery for CRPM. High through-put laboratory techniques for analysing the genetic profile of CRC and CRPM has the power to identify mutation patterns than might predict for treatments and survival outcomes. The results of genetic tests can then be compared to clinical characteristics, such as survival and treatments received. Genes in primary colorectal cancer can be compared to those in CRPM to describe what changes during the metastatic process.

This study will help make progress towards better and personalised treatment options, identifying predictors of treatment success and long-term survival. Improved treatments and better selection of patients may ultimately improve quality of life and help patients live longer.

ELIGIBILITY:
Participants are eligible to be included in the study only if all of the following criteria apply:

1. Patients ≥ 18 years old who have been diagnosed with colorectal cancer and have colorectal peritoneal metastases,
2. have had cytoreductive surgery at the Christie
3. have availability of archival tumour tissue (paired CRC and CRPM)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer peritoneal metastases
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2025-07-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of genetic mutations | 24 months
  Descriptive analysis of the proportion of genetic mutations identified in colorectal cancer and their matched peritoneal metastases: concordance and discordance rates.

SECONDARY OUTCOMES:
Proportion differences of genetic mutations | 24 months
  The descriptive difference in proportion of genetic mutations identified in primary colorectal tumours compared to mutations in colorectal cancer peritoneal metastases. Generate hypotheses about changes that occur during the metastatic process.
Correlations of results | 24 months
  Correlation of results from genetic tests with clinical patient data. Identification of genetic mutations which are associated with differences in survival.
Association with molecular subtypes and categorical variables | 24 months
  Association between molecular subtypes and categorical variables to be measured by Fisher's exact or X2 tests. Associations with continuous variables will be evaluated by Kruskal-Wallis tests or ANOVA. Kaplan-Meier methods will calculate survival outcomes. Univariate and multivariate cox proportional hazard regression models stratified by tumour subtype will identify predictive factors of clinical outcomes. Results with a p-value <0.05 will be considered statistically different.

CONTACTS AND LOCATIONS:
Locations (1):
- Christie Hospital NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided